CLINICAL TRIAL: NCT00003457
Title: Phase II Study Of Antineoplastons A10 And AS2-1 In Patients With Brain Tumors.
Brief Title: Antineoplaston Therapy in Treating Patients With Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066489; BC-BT-9 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-07

CONDITIONS: Refractory Brain Tumors
Keywords: Anaplastic astrocytoma; Anaplastic astrocytoma/Mixed; Astrocytoma; Astrocytoma/Pilocytic; Brainstem glioma; Glioblastoma multiforme; Glioma; Neurocytoma; Primitive neuroectodermal tumor; Tectal glioma
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Glioblastoma; Glioma; Neurocytoma; Neuroectodermal Tumors, Primitive | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with a persistent or recurrent brain tumor will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for adults with persistent or recurrent brain tumors provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of adults with persistent or recurrent brain tumors.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults with persistent or recurrent brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults with persistent or recurrent brain tumors as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in adults with persistent or recurrent brain tumors.

OVERVIEW: This is a single arm, open-label study in which adults with persistent or recurrent brain tumors receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed brain tumor (except brain stem locations) that is unlikely to respond to existing therapy and for which no curative therapy exists
* Evidence of persistent or recurrent brain tumor by MRI scan performed within two weeks prior to study entry
* Tumor must be at least 5 mm
* Ineligible for other Burzynski Research Institute, Inc. brain tumor protocols

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* Hemoglobin at least 9 g/dL
* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed (must be on a stable dose for at least 1 week prior to study entry)

Radiotherapy:

* At least 8 weeks since prior radiotherapy

Surgery:

* Must recover from prior surgery

Other:

* Prior cytodifferentiating agent allowed
* No prior antineoplaston therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1996-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burzynski SR, Janicki TJ, Burzynski GS. A Phase II Study of Antineoplastons A10 and AS2-1 in Adult Patients with Primary Brain Tumors-Final Report (Protocol BT-09). Journal of Cancer Therapy 6(12): 1063-1074, 2015. DOI: 10.4236/jct.2015.612116
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourty patients were recruited between July 1996 and March 2011. All study subjects were seen at the Burzynski Clinic in Houston TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 40
Completed | 31
Not Completed | 9
Not completed — Not evaluable | 9

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: Years] | 36.0 [18.1 to 64.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks; Stable Disease (SD), < 50% decrease and < 25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least 8 weeks; Progressive Disease (PD), >=25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions compared to the lowest sum recorded.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 31
Participants
  Complete Response | 4
  Partial Response | 5
  Stable Disease | 12
  Progressive Disease | 10

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 40
Percentage of participants
  6 months overall survival | 70.0
  12 months overall survival | 50.0
  24 months overall survival | 40.0
  36 months overall survival | 35.0
  48 months overall survival | 30.0
  60 months overall survival | 22.5

ADVERSE EVENTS:
Time Frame: 15 years, 7 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 27/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Hemoglobin (Blood and lymphatic system disorders) | 1 — The Hemoglobin was not related to Antineoplaston therapy.
Cardiac ischemia/infarction (Cardiac disorders) | 1 — The Cardiac ischemia/infarction was not related to Antineoplaston therapy.
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 — The Pericardial effusion (non-malignant) was not related to Antineoplaston therapy.
Central venous catheter infection (General disorders) | 5 — The Central venous catheter infections were not related to Antineoplaston therapy.
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 — The INR (International Normalized Ratio of prothrombin time) was not related to Antineoplaston therapy.
Fatigue (asthenia, lethargy, malaise) Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 — One of the Fatigues (asthenia, lethargy, malaise) was probably related to Antineoplaston therapy.
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 — The Bruising (in absence of Grade 3 or 4 thrombocytopenia) was not related to Antineoplaston therapy.
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 1 — The Pancreatic endocrine: glucose intolerance was not related to Antineoplaston therapy.
Obstruction, GI: Small bowel NOS (Gastrointestinal disorders) | 1 — The Obstruction, GI: Small bowel NOS was not related to Antineoplaston therapy.
Perforation, GI: Duodenum (Gastrointestinal disorders) | 1 — The Perforation, GI: Duodenum was not related to Antineoplaston therapy.
Hemorrhage, CNS (Nervous system disorders) | 2 — The Hemorrhages, CNS were not related to Antineoplaston therapy.
Hemorrhage, GI: Abdomen NOS (Gastrointestinal disorders) | 1 — The Hemorrhage, GI: Abdomen NOS was not related to Antineoplaston therapy.
Infection - Other (Infections and infestations) | 1 — The Infection - Other was not related to Antineoplaston therapy.
Infection (documented clinically): Bladder (urinary) (Renal and urinary disorders) | 1 — The Infection (documented clinically): Bladder (urinary) was not related to Antineoplaston therapy.
Infection (documented clinically): Blood (Infections and infestations) | 5 — The Infections (documented clinically): Blood were not related to Antineoplaston therapy.
Infection (documented clinically): Colon (Infections and infestations) | 1 — The Infection (documented clinically): Colon was not related to Antineoplaston therapy.
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 3 — The Infections (documented clinically): Lung (pneumonias) were not related to Antineoplaston therapy.
Infection (documented clinically): Skin (cellulitis) (Infections and infestations) | 2 — The Infections (documented clinically): Skin (cellulitises) were not related to Antineoplaston therapy.
Lung (pneumonia) (Infections and infestations) | 1 — The Lung (pneumonia) was not related to Antineoplaston therapy.
Hypernatremia (Investigations) | 2 — The Hypernatremias were possibly related to Antineoplaston therapy.
Confusion (Nervous system disorders) | 2 — The Confusions were not related to Antineoplaston therapy.
Neuropathy: motor (Nervous system disorders) | 1 — The Neuropathy: motor was not related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 11 — The Seizures were not related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 — One of the Somnolences/depressed levels of consciousness was possibly related to Antineoplaston therapy.
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 — The Pain: Abdomen NOS was not related to Antineoplaston therapy.
Pain: Pain NOS (General disorders) | 1 — The Pain: Pain NOS was not related to Antineoplaston therapy.
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 — The Dyspnea (shortness of breath) was not related to Antineoplaston therapy.
Flu-like syndrome (Infections and infestations) | 1 — The Flu-like syndrome was not related to Antineoplaston therapy.
Thrombosis/thrombus/embolism (Vascular disorders) | 3 — The Thromboses/thrombi/embolisms were not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 10
Tinnitus (Ear and labyrinth disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 13
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 14
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7
Platelets (Blood and lymphatic system disorders) | 9
Hypertension (Cardiac disorders) | 3
Central venous catheter infection (Infections and infestations) | 13
Non-functional central venous catheter (General disorders) | 13
Central venous catheter - Other (General disorders) | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 28
Fever (General disorders) | 5
Insomnia (General disorders) | 3
Rigors/chills (General disorders) | 7
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 4
Edema/Fluid retention (General disorders) | 15
Anorexia (Gastrointestinal disorders) | 5
Dehydration (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 6
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 16
Hemorrhage, CNS (Nervous system disorders) | 3
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 4
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 7
Infection (documented clinically): Blood (Infections and infestations) | 6
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 4
Infection (documented clinically): Mucosa (Infections and infestations) | 6
Infection (documented clinically): Sinus (Infections and infestations) | 3
Infection (documented clinically): Soft tissue NOS (Infections and infestations) | 3
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 7
Infection (documented clinically): Urinary tract NOS (Infections and infestations) | 5
Opportunistic infection (Infections and infestations) | 5
Albumin, serum-low (hypoalbuminemia) (Investigations) | 5
Alkaline phosphatase (Investigations) | 8
Bicarbonate, serum-low (Investigations) | 4
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 7
Hyperbilirubinemia (Investigations) | 3
Hypercholesteremia (Investigations) | 6
Hyperglycemia (Investigations) | 19
Hypernatremia (Investigations) | 26
Hypertriglyceridemia (Investigations) | 4
Hypocalcemia (Investigations) | 19
Hypoglycemia (Investigations) | 7
Hypokalemia (Investigations) | 37
Hypomagnesemia (Investigations) | 9
Hyponatremia (Investigations) | 3
Hypophosphatemia (Investigations) | 8
Metabolic/Laboratory - Other (Investigations) | 4
Proteinuria (Investigations) | 12
SGOT (Investigations) | 13
SGPT (Investigations) | 14
Uric acid, serum-high (hyperuricemia) (Investigations) | 3
Ataxia (incoordination) (Nervous system disorders) | 5
Confusion (Nervous system disorders) | 14
Dizziness (Nervous system disorders) | 13
Memory impairment (Nervous system disorders) | 6
Mood alteration: Agitation (Nervous system disorders) | 4
Mood alteration: Anxiety (Nervous system disorders) | 3
Mood alteration: Depression (Nervous system disorders) | 4
Neuropathy: motor (Nervous system disorders) | 7
Neuropathy: sensory (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 15
Somnolence/depressed level of consciousness (Nervous system disorders) | 16
Speech impairment (Nervous system disorders) | 10
Tremor (Nervous system disorders) | 5
Vision-blurred vision (Eye disorders) | 7
Pain: Abdomen NOS (Gastrointestinal disorders) | 5
Pain: Back (Musculoskeletal and connective tissue disorders) | 3
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 3
Pain: Head/headache (Nervous system disorders) | 18
Pain: Joint (Musculoskeletal and connective tissue disorders) | 15
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6
Incontinence, urinary (Renal and urinary disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 10
Flu-like syndrome (Infections and infestations) | 5
Thrombosis/thrombus/embolism (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No